CLINICAL TRIAL: NCT02862912
Title: Chloroprocaine Versus Bupivacaine Spinal Anesthesia for Cervical Cerclage
Brief Title: Chloroprocaine Spinal Anesthesia for Cervical Cerclage (CP Spinal)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Richard M. Smiley, Professor of Anesthesiology, Columbia University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Other
Other Study IDs: AAAQ0916
Record Dates: First submitted 2016-08-01; First posted 2016-08-11 (Estimated); Results first posted 2020-05-26 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Adverse Reaction to Spinal Anesthetic; Maternal Care for Cervical Incompetence
Keywords: Chloroprocaine; cervical cerclage; spinal anesthesia; Bupivacaine
MeSH Terms: interventions — chloroprocaine; Bupivacaine; Fentanyl; Sodium Chloride; Fluoridation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloroprocaine (CP) (Experimental): Patients in CP group will receive 3% 2-chloroprocaine 50 mg (1.67 ml) and fentanyl 15 mcg (0.3 ml)
  Interventions: Drug: Chloroprocaine; Drug: Fentanyl
- Bupivacaine (BUP) (Active Comparator): Patients in BUP group will receive hyperbaric 0.75% bupivacaine 9 mg (1.4 ml), with fentanyl 15 mcg (0.3 ml), with saline (0.3 ml) to bring the volume to ~ 2 ml
  Interventions: Drug: Bupivacaine; Drug: Fentanyl; Drug: Saline

INTERVENTIONS:
Drug: Chloroprocaine — Administered as a single injection or continuously through an indwelling catheter - 50 mg
  Other Names: Nesacaine
  Arms: Chloroprocaine (CP)
Drug: Bupivacaine — A dextrose Solution is usually given as an injection - 9 mg (1.4 ml)
  Other Names: Bupivacaine hydrochloride
  Arms: Bupivacaine (BUP)
Drug: Fentanyl — 15 mcg Fentanyl will be included int he spinal anesthetic in both groups
  Other Names: Sublimaze
Drug: Saline — Preservative free normal saline (0.3 ml) to bring the volume to ~ 2 ml
  Other Names: Salt water
  Arms: Bupivacaine (BUP)

SUMMARY:
This study aims to determine whether or not spinal anesthesia with the local anesthetic drug, chloroprocaine, wears off faster than the local anesthetic drug, bupivacaine, and results in faster discharge from the post-anesthesia care unit after surgery.

DETAILED DESCRIPTION:
This will be a prospective, randomized, double blind clinical trial. Subjects will be ASA I and II women ≥18 yrs old with a singleton pregnancy in the 1st or 2nd trimester of pregnancy undergoing cervical cerclage with spinal anesthesia. Patients will be randomly allocated to the chloroprocaine (CP) or bupivacaine group (BUP). Patients will receive spinal anesthesia with either chloroprocaine 50 mg with fentanyl 15 mcg or bupivacaine 9 mg with fentanyl 15 mcg.

Bupivacaine is the most common local anesthetic used for cervical cerclage with spinal anesthesia. Bupivacaine is safe and has been preferred over other medications such as lidocaine, because it is associated with a low incidence of a complication from spinal anesthesia known as "transient neurologic symptoms" - a condition where pain and cramping in the buttocks and lower extremities can be experienced for several days. Bupivacaine is a long-acting local anesthetic agent and therefore has the disadvantage of a prolonged anesthetic recovery that may last a few hours.

Chloroprocaine is a local anesthetic with a fast onset and short duration that may be used for spinal anesthesia for ambulatory procedures. Chloroprocaine is currently used at the research institution for spinal anesthesia for ambulatory surgical patients, especially for lower extremity orthopedic procedures such as knee arthroscopy, as well as for pregnant patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II women
* 18-45 yrs old
* Singleton pregnancy
* Cervical cerclage 1st or 2nd trimester of pregnancy undergoing with spinal anesthesia
* Height 150 - 180 cm
* BMI ≤ 40 kg/m2.

Exclusion Criteria:

* Any contraindication to neuraxial anesthesia (history of neurologic disease (e.g., multiple sclerosis, spinal stenosis, central or peripheral neuropathy)
* Pre-existing/chronic back pain
* Ester local anesthetic allergy, PABA allergy
* History of atypical cholinesterase (CP is metabolized by cholinesterase)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Smiley, MD, Principal Investigator — Columbia University
Locations (1):
- New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A research report will be written and submitted to a peer-reviewed journal
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Submission will be made by December, 2020. Publication availability is to be determined by the peer review process. Once published, the data should be available indefinitely.
Access Criteria: To be determined.

REFERENCES:
- [Background] Camponovo C, Wulf H, Ghisi D, Fanelli A, Riva T, Cristina D, Vassiliou T, Leschka K, Fanelli G. Intrathecal 1% 2-chloroprocaine vs. 0.5% bupivacaine in ambulatory surgery: a prospective, observer-blinded, randomised, controlled trial. Acta Anaesthesiol Scand. 2014 May;58(5):560-6. doi: 10.1111/aas.12291. Epub 2014 Mar 6. PMID 24601887
- [Background] Hejtmanek MR, Pollock JE. Chloroprocaine for spinal anesthesia: a retrospective analysis. Acta Anaesthesiol Scand. 2011 Mar;55(3):267-72. doi: 10.1111/j.1399-6576.2010.02371.x. PMID 21288208
- [Derived] Lee A, Shatil B, Landau R, Menon P, Smiley R. Intrathecal 2-Chloroprocaine 3% Versus Hyperbaric Bupivacaine 0.75% for Cervical Cerclage: A Double-Blind Randomized Controlled Trial. Anesth Analg. 2022 Mar 1;134(3):624-632. doi: 10.1213/ANE.0000000000005653. PMID 34153006

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chloroprocaine (CP) | Bupivacaine (BUP)
Started | 23 | 20
Completed | 22 | 20
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Women with an indication for cervical cerclage with spinal anesthesia
Groups:
- Total: Total of all reporting groups
Arm/Group | Chloroprocaine (CP) | Bupivacaine (BUP) | Total
Number analyzed (Participants) | 23 | 20 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (4) | 34 (6) | 33 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 14 | 12 | 26
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 7 | 21
  White | 7 | 9 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 20 | 43

OUTCOME MEASURES:

1. Primary Outcome: Time to Resolution of Motor Block
Description: The mean difference between groups in time between the end of spinal injection (t IT) to time for no motor block (t motor), i.e. tIT - T motor. Motor block will be assessed using the Bromage scale:
  Bromage Scale I = free movement of the legs and feet = no block II = able to flex knees, with free movement of feet = partial (33%) block III = unable to flex knees, but with free movement of the feet = almost complete (66%) block IV = unable to move legs or feet = complete block (100%)
Time Frame: 3 hours
Population: One protocol violation in the chloroprocaine group led to 22 subjects being analyzed. One block failure in the bupivacaine group led to 19 subjects being analyzed. During analysis it was noted that the motor and sensory block resolution data was missing for 2 subjects in the bupivacaine group so only partial data was available. As a result, 17 participants were analyzed in the bupivacaine group.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Chloroprocaine (CP) | Bupivacaine (BUP)
Number analyzed (Participants) | 22 | 17
minutes | 109 [88 to 148] | 112 [97 to 143]

2. Secondary Outcome: Time to Ambulate
Description: Time from spinal anesthesia placement to ability to ambulate.
Time Frame: 5 hours
Population: One protocol violation in the chloroprocaine group led to 22 subjects being analyzed. One block failure in the bupivacaine group led to 19 subjects being analyzed.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Chloroprocaine (CP) | Bupivacaine (BUP)
Number analyzed (Participants) | 22 | 19
minutes | 158 [137 to 188] | 229 [186 to 332]

3. Secondary Outcome: Time to Void
Description: Time from spinal anesthesia injection to ability to void spontaneously.
Time Frame: 5 hours
Population: In practice, time to void coincided with time to ambulate (to use toilet) and the data is therefore identical to time to ambulate (also time to meet discharge criteria in practice). One protocol violation in the chloroprocaine group led to 22 subjects being analyzed. One block failure in the bupivacaine group led to 19 subjects being analyzed.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Bupivacaine (BUP) | Chloroprocaine (CP)
Number analyzed (Participants) | 19 | 22
minutes | 229 [186 to 332] | 158 [137 to 188]

ADVERSE EVENTS:
Time Frame: Up to postoperative day 1
Arm/Group | Chloroprocaine (CP) | Bupivacaine (BUP)
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 0/23 | 0/20

LIMITATIONS AND CAVEATS:
Despite low dropout risk, we proposed to enroll an additional 4 subjects/group above calculated sample size. The significantly shorter discharge times among some subjects became increasingly apparent. It became untenable to claim clinical equipoise. After the originally calculated sample size was achieved, we decided to stop enrolling new cases, accounting for uneven group numbers. A Shapiro-Wilk test indicated block resolution and discharge time data was non-normal (medians [IQR] reported).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT02862912/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT02862912/Prot_SAP_001.pdf